CLINICAL TRIAL: NCT03831763
Title: Single (Investigator)-Blind, Randomized, Parallel-group Study to Evaluate the Use of Various Assessments of Common Cold Symptoms for Proof of Efficacy of CMS016317
Brief Title: Evaluation of the Use of Various Assessments of Common Cold Symptoms for Proof of Efficacy of ColdZyme Mouth Spray
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Enzymatica AB (Industry)
Collaborators: Analyze & Realize (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 016317
Record Dates: First submitted 2019-01-21; First posted 2019-02-06 (Actual); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Common Cold
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ColdZyme (Active Comparator)
  Interventions: Device: ColdZyme
- Optional care only (No Intervention)

INTERVENTIONS:
Device: ColdZyme — ColdZyme® Mouth Spray is a CE-marked medical device with the following composition: glycerol, water, cod trypsin, ethanol (<1 %), calcium chloride, trometamol and menthol.
  ColdZyme® Mouth Spray consists of a 20 ml bottle, pump, spray nozzle and protective cap.
  Arms: ColdZyme

SUMMARY:
This study evaluates the use of various assessments of common cold symptoms for proof of efficacy of ColdZyme Mouth Spray on naturally acquired common colds. Half of the participants will receive ColdZyme® Mouth Spray while the other half may use optional care as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women
2. Age 18 to 70 years old
3. Increased risk for common cold (at least 3 self-reported occurences of common cold within the last 12 months prior to V1) but generally in good health
4. Readiness to comply with trial procedures:

   * Use of IP as recommended (verum group)
   * Filling in diary
   * Keeping habitual diet and physical activity level
5. Women of child-bearing potential:

   * Have to agree to use appropriate contraception methods
   * Negative pregnancy testing (beta human chorionic gonadotropin test in urine) at V1

Participation is based upon written informed consent by the participant following written and oral information by the investigator regarding nature, purpose, consequences and possible risks of the clinical study.

Exclusion Criteria:

1. Known allergy or hypersensitivity to the components of the investigational product
2. History and/or presence of clinically significant condition/ disorder (self-reported), which per investigator's judgement could interfere with the results of the study or the safety of the subject, e.g.:

   * Nasal disorder (e.g. polyposis, relevant septal deviation, ulcer etc.) and/or reconstructive surgery
   * Acute/chronic airways disease/disorder (e.g. chronic obstructive lung disease, asthma, chronic cough of any origin)
   * Acute psychiatric disorders
   * Any other acute/chronic serious organ or systemic diseases
3. Influenza vaccination within the last 3 months prior to V1 and during the study
4. Regular use of products that may influence the study outcome (e.g. immune suppressants/immune stimulants including natural health products, analgesics/antirheumatics, anti-phlogistics, antitussives/expectorants, mouth or throat therapeutics, decongestants, antibiotics, anti-histaminergic drugs, nasal drops/spray) within the last 4 weeks prior to V1 and during the study (except for the defined optional care)
5. Pregnancy or nursing
6. History of (in the past 12 months prior to V1) or current abuse of drugs, alcohol or medication
7. Participation in the present study of a person living in the same household as the subject
8. Inability to comply with study requirements according to investigator's judgement
9. Participation in another clinical study in the 30 days prior to V1 and during the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2018-01-25 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-05 (Actual)

PRIMARY OUTCOMES:
Difference in the Jackson scale between the study groups | 16+/-4 days from start of common cold symptoms
  Jackson scale - total score, local symptoms, systemic symptoms, 2-item score (sore throat & malaise) as recorded in subject diary twice daily, morning and evening). The Jackson score is calculated by summing the following 8 symptom scores: sore throat, blocked nose, runny nose, cough and sneezing (local symptoms) as well as headache, malaise, and chilliness (systemic symptoms). Symptoms are assessed on a 4-point scale: 0 = none (symptom not present), 1 = mild (sensible, but not disturbing or irritating), 2 = moderate (symptoms sometimes disturbing/irritating), 3 = severe (symptoms disturbing/ irritating most of the time).
Difference in WURSS-21 Quality of Life sub score between the study groups | 16+/-4 days from start of common cold symptoms
  WURSS-21 Quality of Life (QoL) recorded in subject diary once daily, in the evening. WURSS-21 is an evaluative illness-specific quality of life instrument with 21 items, designed to assess the negative impact of acute upper respiratory infection, presumed viral (the common cold). In this study, the QoL part of the WURSS-21 will be applied, from item 12 ("think clearly") to item 20 ("live your personal life").
Difference in the Sore Throat Scale between the study groups | 16+/-4 days from start of common cold symptoms
  The Sore Throat Scale is a 0-10 Likert scale where 0=not sore and 10=very sore. Recorded in subject diary twice daily, morning and evening.
Difference in the Irritated Throat Scale between the study groups | 16+/-4 days from start of common cold symptoms
  Irritated Throat Scale is a 0-10 Likert scale where 0=not irritated and 10=very irritated. Recorded in subject diary twice daily, morning and evening.
Percentage of subjects with prevention of cold outburst | Within 3 days from symptom start
  Based on the assessment of the symptoms recorded in the diary by means of the specified criteria for a common cold episode, as well as the evaluation of any symptoms by the investigator at V2 (whether they are attributable to common cold), the percentage of subjects with prevention of common cold outburst (upon originally having experienced initial symptoms) will be assessed.
Difference in number of findings during physical examination compared between the study groups | From randomisation through study completion, maximum 16 weeks
  Physical examination will be performed using standard products and procedures at all study visits. Physical examination by standard clinical examination of the gastrointestinal tract, cardiovascular system, eyes, respiratory tract, lymph nodes, musculoskeletal system, neurological functions, urogenital tract, thyroid gland and skin.
Blood pressure (mmHg) compared between the study groups | From randomisation through study completion, maximum 16 weeks
  Sitting blood pressure (mmHg), systolic and diastolic, will be measured using standard products and procedures at all study visits.
Pulse rate (bpm) compared between the study groups | From randomisation through study completion, maximum 16 weeks
  Pulse rate (bpm) will be measured using standard products and procedures at all study visits.
Number of subjects with adverse events | From randomisation through study completion, maximum 16 weeks
  Any AE that occurs during the course of the study.
Number of device deficiencies | During IP use, maximum 12 days from symptom start
  Device deficiencies occurring in the active group (verum)

OTHER OUTCOMES:
Duration of common cold symptoms | 16+/-4 days from start of common cold symptoms
  Number of days since start of cold symptoms until the end of the symptoms (defined as the last day with one or more symptoms followed by at least two symptom-free days (subjects have to answer "No" to the question "Do you think that you are still sick with this respiratory infection?" for 2 days in a row)).
Use of concomitant treatment/remedies | 16+/-4 days from start of common cold symptoms
  Use of any concomitant treatment/remedies, reported in subject diary once daily, in the evening
Global evaluation of efficacy by subjects at study end | 16+/-4 days from start of common cold symptoms
  The subjects in the verum group will evaluate the efficacy of the IP (global scaled evaluation with "very good", "good", "moderate" and "poor") at study end.

CONTACTS AND LOCATIONS:
Overall Officials: Ralf Uebelhack, Prof. MD, Principal Investigator — analyze & realize GmbH
Locations (7):
- Germany (7):
  - analyze & realize GmbH, Berlin
  - Barbara Grube, Berlin
  - Dr. med. Petra Sandow and Eugenia Fischkina, Berlin
  - Dr. med. Ruhland, Berlin
  - Klinische Forschung Berlin, Berlin
  - POLIKUM Institut GmbH, Berlin
  - Thomas Wünsche, Berlin

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported, after deidentification (text, tables, figures and appendices) will be shared with researchers who provide a methodologically sound proposal, to achieve aims in hte approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Individual participant data that underlie the results reported, after deidentification (text, tables, figures and appendices) will be shared with researchers who provide a methodologically sound proposal, to achieve aims in hte approved proposal. Proposals should be directed to fredrik.lindberg@enzymatica.com. To gain access, data requestors will need to signa data access agreement.